CLINICAL TRIAL: NCT02923362
Title: Registry of Outcomes From AntiReflux Surgery (ROARS)
Brief Title: Registry of Outcomes From AntiReflux Surgery
Acronym: ROARS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: The Heartburn Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: THF001
Record Dates: First submitted 2016-10-03; First posted 2016-10-04 (Estimated); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Gastroesophageal Reflux Disease; Hiatal Hernia
Keywords: GERD; Reflux; Acid Reflux; Heartburn; Regurgitation; Laryngopharyngeal Reflux; Hiatal Hernia; LPR; LINX; Magnetic Sphincter Augmentation; Antireflux Surgery; Nissen
MeSH Terms: conditions — Gastroesophageal Reflux; Hernia, Hiatal; Heartburn; Laryngopharyngeal Reflux | interventions — Fundoplication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Laparoscopic Fundoplication Group: This group of patients are surgical candidates based on preoperative testing results for laparoscopic fundoplication antireflux procedure and possible hiatal hernia repair.
  Interventions: Procedure: Laparoscopic Fundoplication
- LINX Antireflux Device Group: This group of patients are surgical candidates based on preoperative testing results for the laparoscopic LINX antireflux device placement and possible hiatal hernia repair.
  Interventions: Device: LINX Antireflux

INTERVENTIONS:
Procedure: Laparoscopic Fundoplication — The gastric fundus of the stomach is wrapped or plicated around the lower end of the esophagus and and stitched in place reinforcing the closing function of the lower esophageal sphincter. The hiatus is also narrowed down with sutures or mesh to prevent or treat a concurrent hiatal hernia.
  Other Names: Nissen Fundoplication; Fundoplication; Fundoplasty; Hiatal Hernia Repair; Partial Fundoplication
  Groups: Laparoscopic Fundoplication Group
Device: LINX Antireflux — The LINX is a flexible band of interlocked titanium beads with a magnetic core. The LINX is placed around the lower esophageal sphincter to help restore the function of the LES by preventing reflux into the esophagus.
  Other Names: LINX System; LINX Implant; LINX Reflux Management System; LINX Magnetic Sphincter Augmentation
  Groups: LINX Antireflux Device Group

SUMMARY:
Prospective registry comparing outcomes after laparoscopic treatment of gastroesophageal reflux disease and hiatal hernia.

DETAILED DESCRIPTION:
This is a prospective, multi center, observational database of patients that are having surgical laparoscopic antireflux procedure and/or hiatal hernia repair, including laparoscopic Nissen fundoplication and Magnetic Sphincter Augmentation with the LINX device. Patients meeting registry inclusion and exclusion will be followed for 5 years with standardized quality of life surveys and appropriate standard of care testing. Up to 40 sites will participate with total enrollment of 1000 patients.

The main objectives are to collect data from everyday clinical practices and track patients from preoperative assessments to 5 years post surgical intervention to evaluate symptoms, medication use and side effects.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be at least 21years of age and at least the minimum Age of Majority according to applicable state law.
* Subject is a suitable surgical candidate, i.e. is able to undergo appropriate anesthesia and endoscopic procedure or laparoscopic surgery.
* Appropriate indications for and documentation of disease process requiring surgery. (Documented gastroesophageal reflux disease by accepted endoscopic or ambulatory reflux monitoring criteria, or have a hiatal hernia that meets accepted criteria for repair (e.g. large paraesophageal hernia with chest pain)).
* Subject is willing and able to cooperate with follow-up examinations
* Subject has been informed of the study procedures and treatment and has signed an informed consent for the study.

Exclusion Criteria:

* Suspected or confirmed esophageal or gastric cancer.
* Cannot understand trial requirements or is unable to comply with follow-up schedule
* Pregnant or nursing, or plans to become pregnant during the course of the study
* Medical illness (i.e. congestive heart failure) that may cause the subject to be non-compliant with or able to meet the protocol requirements or is associated with limited life expectancy (i.e. less than 3 years)
* Diagnosed psychiatric disorder (e.g. bipolar, schizophrenia, etc.), subjects that exhibit depression that are on appropriate medication(s) are allowable.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patient over the age of 21 with no maximum age who meet the eligibility for anti reflux and or hiatal hernia repair surgery
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2016-05; Primary Completion 2023-03 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Quality of Life reported by patient | 5 Years
  Standard GERD Quality of Life Assessment

CONTACTS AND LOCATIONS:
Overall Officials: Reginald Bell, MD, Principal Investigator — The Heartburn Foundation
Locations (19):
- United States (19):
  - Advanced Surgeons, PC, Birmingham, Alabama
  - University of Southern Alabama, Mobile, Alabama
  - The Arkansas Heartburn Treatment Center, Heber Springs, Arkansas
  - Bass Medical Group, Walnut Creek, California
  - HealthOne Cardiothoracic Surgery Associates, Aurora, Colorado
  - Institute of Esophageal and Reflux Surgery, Englewood, Colorado
  - Suncoast Surgical Associates, Brandon, Florida
  - South Florida Surgical Specialists, LLC, Coral Springs, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Tampa Bay Reflux Center, Riverview, Florida
  - The Tampa Bay Reflux Center, Tampa, Florida
  - Coastal Carolina Bariatric and Surgical Center, Summerville, South Carolina
  - Baylor Scott and White Research Institute, Dallas, Texas
  - Baylor University Medical Center at Dallas, Dallas, Texas
  - Houston Methodist Research Institute, Houston, Texas
  - North Texas Surgical Oncology Associates, Plano, Texas
  - Swedish Health Services, Seattle, Washington
  - Affinity Medical Group, Chilton, Wisconsin
  - Froedtert & The Medical College of Wisconsin Hospitals and Health Partners, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No